CLINICAL TRIAL: NCT03847311
Title: Double Blind Trial Investigating the Role of Sulfasalazine in Decreasing Opioids Requirements in Breast Cancer Patients
Brief Title: Sulfasalazine in Decreasing Opioids Requirements in Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mohab Ibrahim, PhD MD, Director, Comprehensive Pain Management Clinic Associate Professor, Anesthesiology, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1605576856; 5R21CA245411-02 (NIH)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Chronic Pain Due to Malignancy (Finding)
MeSH Terms: conditions — Breast Neoplasms; Signs and Symptoms | interventions — Sulfasalazine

STUDY DESIGN:
Intervention Model Description: Double blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The research pharmacist will randomize and prepare the drugs so that the drugs look similar, the pharmacist will dispense the drugs into vials, and label the drug so is not identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebos (Placebo Comparator): Subjects will receive sugar pill.
  Interventions: Drug: Placebos
- Sulfasalazine (Active Comparator): Subjects will receive the active drug.
  Interventions: Drug: Sulfasalazine

INTERVENTIONS:
Drug: Sulfasalazine — This group will receive supplies for 3 months of sulfasalazine at an initial dose of 0.5 gram three times a day for a week then at a dose of 1 gram three times a day for the remainder of the 3 months. Subjects will be asked to take their medications with every meal in addition to their regular pain medications.
  Other Names: Active treatment
  Arms: Sulfasalazine
Drug: Placebos — This group will receive supplies for 3 months of sugar pills three times a day for 3 months. Subjects will be asked to take their medications with every meal in addition to their regular pain medications.
  Other Names: Non-active
  Arms: Placebos

SUMMARY:
Cancer in general, and breast cancer in specific, is a significant health problem in the USA and the rest of the world. With the improvement of new surgical approaches and chemotherapies to manage breast cancer, the number of patients with breast cancer are now living longer. This great achievement created an unexpected problem. For some breast cancer patients, with bone metastases, the pain is worse than the cancer. The golden standard to manage pain is opioids. Patients with cancer-induced bone pain are now taking increasing doses of opioids to control their pain. Sadly, opioids come with significant side effects that limit the amount of opioids that can be safely given. Many attempts have been tried to create better regiments for pain control to lower the need for opioids. There has not been significant success in that area. A better approach would be to add a non-opioid agent that has dual mechanisms of action. This may create synergism to better control pain while lowering the doses of opioids needed and lowering side effects. Sulfasalazine poses such quality it is a safe anti-inflammatory drug with established safety profile. It has been in use for over 50 years for the treatment of inflammatory conditions such as arthritis. In addition to its anti-inflammatory characteristics, sulfasalazine has the capacity to decrease the survival of cancer cells, also to lower the number of inflammatory mediators released by cancer cells. In short, sulfasalazine inhibit the influx of cysteine into cancer cells and the efflux of glutamate. Cysteine is needed for cell survival against oxidative stress, while glutamate activate pain receptors. Therefore, sulfasalazine will act as anti-inflammatory, an agent to accelerate cancer cells death and decreasing the released glutamate which activate pain receptors. This one agent with 3 mechanisms of actions may lower the amount of opioid needed for these patients while maintaining or improving their pain. Lowering of opioid dosing may also improve the side effects associated with opioid use. The purpose of this trial is to co-administer sulfasalazine with opioids to cancer patients and characterize their pain and the opioid use. Our hypothesis is that adding sulfasalazine to the pain medication, will lower the amount of opioids used and lower the side effects. This may improve the quality of life for patients and decrease the risks of using high amount of opioids for the patients, their families, and society in general.

DETAILED DESCRIPTION:
In the United States, approximately one in two men and one in three women will develop cancer. Today, more than 15 million people live with cancer in the United States alone. The direct annual medical cost of cancer is over 86 billion US dollars. The indirect cost, representing loss of wages and productivity, exceeds 130 billion US dollars annually. It is estimated that 90% of all cancer patients report pain. About 63% of patients with advanced stage cancer or with metastasis suffer from pain that is classified as "moderate to severe". The majority of cancer patients suffer from excruciating pain. Even those who survive cancer may still experience pain. Of all cancer survivors, 59% report pain secondary to chemotherapy. Even after patients are cured from their cancer, 33% of these patients will still suffer from severe pain due to their chemotherapy. Inadequate pain management results in 67% of patients with severe pain. Notably, 32% of cancer patients reported a desire for suicide secondary to their pain.

Opioids have been the gold standard to treat cancer pain. Sadly, there are many side effects associated with chronic opioid use. It has been shown in animal models that chronic use of opioids has been associated with paradoxical effects. Rats that have been exposed to chronic opioids developed hyperalgesia, which is an exaggerated response to a painful stimulus and allodynia, which is a painful response to a non-painful stimulus. There have been several mechanisms proposed to explain the paradoxical hyperalgesia phenomena observed. This phenomenon has been recognized in patients inflected with chronic pain and managed with chronic opioid. It has been long observed that patients with chronic pain require gradually increasing doses of opioids. The reasons for this increase in opioid requirement may be complicated. While the progression of the disease may play a significant part in increasing doses of opioid, other factors such as tolerance and opioid induced hyperalgesia cannot be ignored. Tolerance is a characteristic of opioids that is well investigated and results in increasing the doses of opioids to maintain the original analgesic effects. Changing of brain circuitry enables opioids to play a sinister role allowing it to produce pain. Additionally, patients develop physical dependence with their use of opioids. A more significant aspect of chronic use of opioid is the psychological dependence on opioids. While its understandable and necessary for cancer patients to have opioids to control their pain, finding adjuvant pain control therapy may lessen the amount of opioids needed. Using neuropathic pain medications as adjuvants to supplement opioids had mixed results. Therefore, a different agent with different mechanism is action may be needed for better pain control with less opioids.

Cancer cells have high metabolic rate that generate high oxidative stress burden. Cancer cells require glutathione to combat oxidative stress for survival. Cysteine is required for the synthesis of glutathione. Cells acquire cysteine be exchanging intracellular glutamate for the extra cellular cysteine through the Cysteine/Glutamate antiporter. Excreting glutamate results in increased pain through the activation of N-methyl-D-aspartate receptor (NMDA). If an agent can be identified that inhibits the Cysteine/Glutamate antiporter, the cancer cells will have less chances of survival secondary to decreased glutathione that's is needed for protection from oxidative stress. Additionally, decreased amount of the glutamate secreted from the cells may lower the amount of pain produced.

Sulfasalazine is a safe and well-established anti-inflammatory drug with potent inhibitory properties of the cysteine/glutamate antiporter. Utilizing sulfasalazine for cancer patients, in conjunction with opioids, may reduce the amount of opioids needed in two different methods. First, sulfasalazine may decrease the survival rate of cancer cells, thus lowering the mechanical burden of the cancer. Second, sulfasalazine may decrease the amount of glutamate released by cancer cell resulting in less activation of the NMDA receptor.

The investigator proposes a clinical trial to administer sulfasalazine to initially focus on breast cancer patients with pain. The pain may be from the primary tumor or from metastasis. The investigator hypothesis that sulfasalazine will reduce cancer pain, the amount of the opioids needed, and the undesirable side effects associated with high doses of opioid.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient age 18 - <95 years old capable of understanding and providing consent in English and capable of complying with the outcome used.
* Diagnosis of cancer with pain moderate to severe pain on stable doses of opioids
* 3-day average numeric pain rating score (NPRS) for pain of at least 5/10 at baseline evaluation.
* Patient consents to double blind design of the experiment in a shared decision- making process with the treating physician.
* Pain duration of at least 6 weeks or more.
* Prognosis greater than 6 months.
* Able to take oral medication

Exclusion Criteria:

* Those receiving remuneration for their pain treatment (e.g., disability, worker's compensation).
* Those involved in active litigation relevant to their pain.
* Subjects with intestinal or urinary obstruction or at risk of such disorders.
* Porphyria
* Blood dyscrasias, hepatic or renal disease.
* Taking medications that may interact with sulfasalazine.
* Taking Lapatinib or Digoxin.
* No sustained hypercalcemia.
* Hypersensitivity to sulfasalazine, its metabolites, sulfonamides, or salicylates.
* The Subject is incarcerated.
* Those unable to read English and complete the assignment in English.
* Addictive behavior, severe clinical depression, or psychotic features.
* Possible pregnancy or lactation.

Ages: 18 Years to 94 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohab M Ibrahim, PhD., MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Banner University Medical Center South, Tucson, Arizona
  - Banner University Medical Center North Campus, Tucson, Arizona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lifetime Probability of Developing and Dying From Cancer for 23 sites, 2009-2011. 2014.
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Carinci AJ, Mao J. Pain and opioid addiction: what is the connection? Curr Pain Headache Rep. 2010 Feb;14(1):17-21. doi: 10.1007/s11916-009-0086-x. PMID 20425210
- [Background] Starrels JL, Becker WC, Alford DP, Kapoor A, Williams AR, Turner BJ. Systematic review: treatment agreements and urine drug testing to reduce opioid misuse in patients with chronic pain. Ann Intern Med. 2010 Jun 1;152(11):712-20. doi: 10.7326/0003-4819-152-11-201006010-00004. PMID 20513829
- [Background] Bekhit MH. Opioid-induced hyperalgesia and tolerance. Am J Ther. 2010 Sep-Oct;17(5):498-510. doi: 10.1097/MJT.0b013e3181ed83a0. PMID 20844348
- [Background] Lee M, Silverman SM, Hansen H, Patel VB, Manchikanti L. A comprehensive review of opioid-induced hyperalgesia. Pain Physician. 2011 Mar-Apr;14(2):145-61. PMID 21412369
- [Background] Mao J, Sung B, Ji RR, Lim G. Chronic morphine induces downregulation of spinal glutamate transporters: implications in morphine tolerance and abnormal pain sensitivity. J Neurosci. 2002 Sep 15;22(18):8312-23. doi: 10.1523/JNEUROSCI.22-18-08312.2002. PMID 12223586
- [Background] Vanderah TW, Suenaga NM, Ossipov MH, Malan TP Jr, Lai J, Porreca F. Tonic descending facilitation from the rostral ventromedial medulla mediates opioid-induced abnormal pain and antinociceptive tolerance. J Neurosci. 2001 Jan 1;21(1):279-86. doi: 10.1523/JNEUROSCI.21-01-00279.2001. PMID 11150345
- [Background] Arner S, Rawal N, Gustafsson LL. Clinical experience of long-term treatment with epidural and intrathecal opioids--a nationwide survey. Acta Anaesthesiol Scand. 1988 Apr;32(3):253-9. doi: 10.1111/j.1399-6576.1988.tb02725.x. PMID 3364150
- [Background] Williams JT, Ingram SL, Henderson G, Chavkin C, von Zastrow M, Schulz S, Koch T, Evans CJ, Christie MJ. Regulation of mu-opioid receptors: desensitization, phosphorylation, internalization, and tolerance. Pharmacol Rev. 2013 Jan 15;65(1):223-54. doi: 10.1124/pr.112.005942. Print 2013 Jan. PMID 23321159
- [Background] Ballantyne JC, Mao J. Opioid therapy for chronic pain. N Engl J Med. 2003 Nov 13;349(20):1943-53. doi: 10.1056/NEJMra025411. No abstract available. PMID 14614170
- [Background] Bar Ad V. Gabapentin for the treatment of cancer-related pain syndromes. Rev Recent Clin Trials. 2010 Sep;5(3):174-8. doi: 10.2174/157488710792007310. PMID 20482492
- [Background] Takahashi H, Shimoyama N. A prospective open-label trial of gabapentin as an adjuvant analgesic with opioids for Japanese patients with neuropathic cancer pain. Int J Clin Oncol. 2010 Feb;15(1):46-51. doi: 10.1007/s10147-009-0009-1. PMID 20072794
- [Background] Estrela JM, Ortega A, Obrador E. Glutathione in cancer biology and therapy. Crit Rev Clin Lab Sci. 2006;43(2):143-81. doi: 10.1080/10408360500523878. PMID 16517421
- [Background] Griffith OW. Biologic and pharmacologic regulation of mammalian glutathione synthesis. Free Radic Biol Med. 1999 Nov;27(9-10):922-35. doi: 10.1016/s0891-5849(99)00176-8. PMID 10569625
- [Background] Lo M, Wang YZ, Gout PW. The x(c)- cystine/glutamate antiporter: a potential target for therapy of cancer and other diseases. J Cell Physiol. 2008 Jun;215(3):593-602. doi: 10.1002/jcp.21366. PMID 18181196
- [Background] Gout PW, Buckley AR, Simms CR, Bruchovsky N. Sulfasalazine, a potent suppressor of lymphoma growth by inhibition of the x(c)- cystine transporter: a new action for an old drug. Leukemia. 2001 Oct;15(10):1633-40. doi: 10.1038/sj.leu.2402238. PMID 11587223
- [Background] Klotz U. Clinical pharmacokinetics of sulphasalazine, its metabolites and other prodrugs of 5-aminosalicylic acid. Clin Pharmacokinet. 1985 Jul-Aug;10(4):285-302. doi: 10.2165/00003088-198510040-00001. PMID 2864155
- [Derived] Wang F, Oudaert I, Tu C, Maes A, Van der Vreken A, Vlummens P, De Bruyne E, De Veirman K, Wang Y, Fan R, Massie A, Vanderkerken K, Shang P, Menu E. System Xc- inhibition blocks bone marrow-multiple myeloma exosomal crosstalk, thereby countering bortezomib resistance. Cancer Lett. 2022 Jun 1;535:215649. doi: 10.1016/j.canlet.2022.215649. Epub 2022 Mar 18. PMID 35315341

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebos | Sulfasalazine
Started | 3 | 4
Completed | 2 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebos | Sulfasalazine | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (8.0) | 69.5 (4.6) | 65.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Pain Relief.
Description: Brief Pain Inventory (BPI) pain severity score. Scale range: 0 (no pain) to 10 (worst pain imaginable) Higher values represent a worse outcome.
Time Frame: Twelve weeks
Population: All subjects who completed study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebos | Sulfasalazine
Number analyzed (Participants) | 2 | 3
score on a scale | 1.9 (0.2) | 0.5 (0.4)

2. Secondary Outcome: Decrease Opiate Dose.
Description: Morphine Milligram Equivalents (MME) per day at 12 weeks.
Time Frame: Twelve weeks
Population: All subjects who completed the study.
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents per day
Arm/Group | Placebos | Sulfasalazine
Number analyzed (Participants) | 2 | 4
Morphine Milligram Equivalents per day | 39.4 (14.3) | 33.2 (38.2)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 12 weeks
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the clinicaltrials.gov definitions.
Arm/Group | Placebos | Sulfasalazine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebos (N=3) | Sulfasalazine (N=4)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0 (0) — General Disorders and administration site conditions
Fatigue (General disorders) | 1 (1) | 0 (0) — General Disorders and administration site conditions
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) — General Disorders and administration site conditions
Pain (General disorders) | 0 (0) | 1 (1) — General Disorders and administration site conditions
Urinary Tract Infection (Infections and infestations) | 1 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2)
White blood cell decreased (Investigations) | 2 (10) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (7) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (6) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT03847311/Prot_002.pdf
  • Informed Consent Form (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT03847311/ICF_001.pdf